CLINICAL TRIAL: NCT06677229
Title: Phase 1b/2a Clinical Trial in Early Acute Spinal Cord Injury (SCI): a Single Blinded, Randomized, Proof-of-Concept Study to Determine the Safety, Tolerability and Efficacy of TZ-161
Brief Title: Phase 1b/2a Clinical Trial to Determine the Safety, Tolerability and Efficacy of TZ-161 in Spinal Cord Injury
Acronym: eSpine
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Technophage, SA (Industry)
Collaborators: VectorB2B (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TZ-161-101; 2023-509207-33-01 (EU CTIS Number)
Record Dates: First submitted 2024-11-04; First posted 2024-11-06 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Acute Spinal Cord Injury (SCI)
Keywords: acute spinal cord injury; TZ-161; Eletriptan Hydrobromide; Eletriptan HBr; serotonin receptor; 5-HT receptor; Relert; Relpax
MeSH Terms: interventions — eletriptan

STUDY DESIGN:
Masking Description: Although this clinical trial is an open label study for both study subjects and site personnel, in order to minimise bias, the study will employ the use of blinded raters for performing the following efficacy-related endpoints/tests, hence the denomination of single-blinded study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Arm Randomized to IMP (Eletriptan HBr) + SOC (Experimental)
  Interventions: Drug: Eletriptan HBr 40 mg
- Control Arm after SCI Randomized to SOC (No Intervention)

INTERVENTIONS:
Drug: Eletriptan HBr 40 mg — Oral administration of Eletriptan HBr in the form of tablets, 40 mg once daily (q.d.) for a total of 6 days, together with their usual SOC treatment.
  Arms: Experimental Arm Randomized to IMP (Eletriptan HBr) + SOC

SUMMARY:
Technophage identified a promising compound, Eletriptan hydrobromide, that intends to use as a repurposed drug, for the treatment of acute spinal cord injury (SCI) in human subjects. Eletriptan hydrobromide is a well characterized molecule, that has been clinically available for over two decades for the treatment of migraines. It presents a good and manageable safety profile, including for the regimen selected for this trial, and it is generally well tolerated, with minimal side effects. This is an important consideration to have when using repurposed drugs for the treatment of other indications. Technophage believes that the preclinical data collected, in combination with the acceptable safety profile of Eletriptan hydrobromide, support its use as a repurposed drug for the treatment of SCI in humans.

DETAILED DESCRIPTION:
Eletriptan hydrobromide (HBr) is a second-generation serotonin (5-HT) receptor agonist with high affinity for 5-HT1B, 5-HT1D and 5-HT1F receptors approved for the acute treatment of the headache phase of migraine attacks, with or without aura. 5-HT is a monoamine neurotransmitter synthesized in several subpopulations of brainstem neurons and plays an important role in vertebrate locomotion. Following spinal cord injury (SCI) there is a disruption of descending serotonergic projections to spinal motor areas, which results in a subsequent 5-HT depletion, 5-HT transporter dysregulation, as well as elevated expression, hyper-sensitivity and/or constitutive auto-activation of specific 5-HT receptors. Technophage identified a new possible therapeutic indication for Eletriptan HBr, showing its locomotor recovery properties in two different animal models of injury. Based on preclinical findings, Technophage intends to test Eletriptan HBr in the clinical environment, as a repurposed drug, for the treatment of acute SCI in human subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 18-65 years old.
2. Subjects with clinical diagnosis of acute SCI that comply with the following:

   1. Injury located on the thoracic region (T1 to T12).
   2. With clinical suspicion of a single traumatic (contusion) lesion.
   3. AIS grade of grade B, C or D with a motor score less than or equal to 3 in at least one key muscle of a lower limb.
   4. Ability to perform injury-to-drug administration ≤ 24 hours after SCI.
3. Subjects willing and able to provide an informed consent.
4. Subjects willing and able to complete the study and comply with instructions. The use of Relert in the elderly is not recommended, due to the fact that the safety and effectiveness of Eletriptan HBr in patients over 65 years of age had not been systematically evaluated, as a consequence of the small number of patients in this age group in clinical trials.

Exclusion Criteria:

1. Clinical or imaging suspicion of multi-lesion or extra-thoracic contusions on diagnostic CT scan and on MRI at 48H*.
2. Subjects in coma or with significant cognitive impairment in the opinion of the investigator.
3. Subjects presenting mechanical ventilation dependence.
4. Subjects with past medical history of any - structural - neurological disorder of the central or peripheral nervous system, including past spinal cord injury. Furthermore, subjects with spine/bone-related medical history (prior to SCI) that in the opinion of the investigator are not yet resolved or previous lesions that are located in the same area of the study SCI should also be excluded.
5. Subjects with dysphagia or inability to swallow tablets.
6. Women who are breastfeeding or who are pregnant. Pregnancy to be excluded during screening by presence of a negative blood pregnancy test.
7. Subjects with active malignancy, or malignancy in the last 5 years if subject is currently undergoing treatment with prohibited medication.
8. Subjects that have recently used Eletriptan HBr (within the last 24h).
9. Subjects presenting clinically significant ECG abnormalities (Wolff-Parkinson-White syndrome or arrhythmias associated with other cardiac accessory conduction pathway disorders) at screening.
10. Subjects presenting any contraindications, special warnings, and precautions regarding IMP administration, as per described in the SmPC of Eletriptan HBr:

    1. Ischemic CAD, such as angina pectoris, history of myocardial infarction, and documented silent ischemia, or coronary artery vasospasm, including Prinzmetal's angina.
    2. Wolff-Parkinson-White syndrome or arrhythmias associated with other cardiac accessory conduction pathway disorders.
    3. History of stroke, TIA, or history or current evidence of hemiplegic or basilar migraine because these patients are at a higher risk of stroke.
    4. Peripheral vascular disease.
    5. Ischemic bowel disease.
    6. Uncontrolled hypertension.
    7. Recent use (i.e., within 24 hours) of serotonin receptor agonists
    8. Coadministration with SSRIs, SNRIs, TCAs, and MAO due to risk of serotonin syndrome.
    9. Recent use (i.e., within 24 hours) of drugs containing ergotamine or ergot-like substances (such as dihydroergotamine or methysergide)
    10. Hypersensitivity to IMP and its excipients (angioedema and anaphylaxis seen).
11. The following medications and/or substances are not allowed due to potential interaction with Eletriptan HBr or inhibition of the CYP3A4 system (recent use, i.e., within at least 72 hours):

    1. Cimetidine; ketoconazole; itraconazole; fluconazole, erythromycin; clarithromycin, troleandomycin, verapamil, and MAO inhibitors [such as isocarboxazid (Marplan), phenelzine sulfate (Nardil), tranylcypromine (Parmate), selegiline (Emsam)], pioglitazone, and valerian.
    2. Antiretrovirals - such as ritonavir, indinavir, nelfinavir, efavirenz and nevirapine.
    3. Other prohibited concomitant medications include haloperidol, trazodone, triazolam, nefazodone, diltiazem, carbamazepine, phenytoin, oxcarbazepine, and phenobarbital.
    4. St. John's Wort (Hypericum perforatum).
12. Subjects with known liver disease (except for Child Pugh A) or severe hepatic impairment.
13. Subjects with known renal disease or severe renal impairment - exclude if eGFR below 50 ml/min.
14. Subjects that have participated in any other study in the last 3 months or plan to participate in another study at any time during this clinical trial.
15. Subjects that have foreign magnetic metal bodies or other conditions that render them unable to perform MRI.
16. Any other issue that, in the opinion of the investigator, makes the subject unsuitable for study participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Adverse effects | Between Day 1 and Month 6 in IMP plus SOC compared to SOC alone
  Incidence of treatment-emergent AEs and treatment-emergent SAEs

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario La Paz, Madrid

IPD SHARING:
Plan to Share IPD: No